CLINICAL TRIAL: NCT03191331
Title: Intervention Study on Dietary Changes in Relation to Weight Gain and Prevalence of Gestational Diabetes During Pregnancy
Brief Title: Dietary Intervention, Gestational Weight Gain and Gestational Diabetes.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Eastern Finland (Other)
Responsible Party: Principal Investigator, Reeta Lamminpää, post doctoral researcher, University of Eastern Finland
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: Dietary intervention1619
Record Dates: First submitted 2017-05-29; First posted 2017-06-19 (Actual); Last update posted 2020-03-27 (Actual); Status verified 2020-03

CONDITIONS: Dietary Habits; Gestational Diabetes; Weight Gain; Overweight and Obesity
Keywords: dietary intervention; gestational weight gain; gestational diabetes; overweight; obesity
MeSH Terms: conditions — Feeding Behavior; Diabetes, Gestational; Weight Gain; Overweight; Obesity; Gestational Weight Gain | interventions — Diet Therapy

STUDY DESIGN:
Intervention Model Description: intervention group and control group.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Experimental): Dietary intervention. Intervention group will receive written material on healthy diet during pregnancy, nutritional guidance given by public health nurses at each maternity care clinic visit and group meeting with dietician x2.
  Interventions: Behavioral: Dietary intervention
- Control group (No Intervention): The control group will receive written material on healthy diet during pregnancy, otherwise basic care and guidance at maternity care clinics.

INTERVENTIONS:
Behavioral: Dietary intervention — Written material on healthy diet during pregnancy, dietary counseling at each maternity clinic visit given by public health nurse, group meeting with a dietician x2.
  Arms: Intervention group

SUMMARY:
The aim of this pilot study is to conduct a dietary intervention for overweight (body maas index BMI≥25) and obese (BMI≥30) pregnant women in two maternity care clinics and explore the effect of the intervention on gestational weight gain and the prevalence of gestational diabetes between the intervention and control groups.

DETAILED DESCRIPTION:
Half of the women are allocated to the intervention group and another half for the control group. The intervention group will get written material of healthy diet during pregnancy as well as emphasized nutritional guidance given by public health nurses at each visit in the maternity care clinic. There will also be two group meetings with a dietitian. The control group will get the same written material, but otherwise basic care and guidance at each visit in the maternity care clinics. The collected data of both groups include the information on weight gain, the result of an oral glucose tolerance test and 4 day food records, Three factor eating questionnaire (TFEQ R-18) and Binge Eating Scale (BES).

ELIGIBILITY:
Inclusion Criteria:

* Age less than 35 years
* BMI 25 or over
* healthy, no chronic medical conditions
* singleton pregnancy
* first trimester of pregnancy at the time of recruitment

Exclusion Criteria:

* Age 35 and older
* BMI less than 25
* chronic medical conditions
* multiple pregnancy
* pregnancy at second or third trimester at the time of recruitment

Ages: 18 Years to 35 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Eligibility is based on gender
Enrollment: 13 (Actual)
Dates: Start 2017-06-06 (Actual); Primary Completion 2019-06-01 (Actual); Study Completion 2019-06-01 (Actual)

PRIMARY OUTCOMES:
gestational weight gain (GWG) | from first to third trimester of pregnancy, gestational weeks
  gestational weight gain from 1st trimester of pregnancy until childbirth, measured at each maternity clinic visit

SECONDARY OUTCOMES:
gestational diabetes mellitus (GDM), | gestational weeks 12-16
  GDM is measured by the result of an oral glucose tolerance test (OGTT)
eating habits | 1st, 2nd and 3rd trimester of pregnancy, gestational weeks
  eating habits are measured by 4 day food records
eating habits | 1st, 2nd and 3rd trimester, gestational weeks
  Eating habits are measured by TFEQ R-18 questionnaire
Eating habits | 1st, 2nd and 3rd trimester, gestational weeks
  Eating habits are measured by Binge Eating Scale (BES)

CONTACTS AND LOCATIONS:
Overall Officials: Reeta Lamminpää, PhD, Principal Investigator — University of Eastern Finland, Department of Nursing Science
Locations (2):
- Finland (2):
  - Neulamäki antenatal care clinic, Kuopio
  - Pyörö antenatal care clinic, Kuopio

IPD SHARING:
Plan to Share IPD: No